CLINICAL TRIAL: NCT03327792
Title: A Pilot Study on the Safety and Efficacy of Mavoglurant in Alcohol Drinking
Brief Title: Mavoglurant in Alcohol Drinking
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Suchitra Krishnan-Sarin, Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2000021703; 2P50AA012870-21 (NIH)
Record Dates: First submitted 2017-10-27; First posted 2017-10-31 (Actual); Results first posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Alcohol Drinking
MeSH Terms: conditions — Alcohol Drinking | interventions — mavoglurant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 200 mg Mavoglurant (Experimental): 200 mg mavoglurant once daily for 7-10 days
  Interventions: Drug: Mavoglurant
- Placebo (Placebo Comparator): Placebo once daily for 7-10 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mavoglurant — 200 mg Mavoglurant
  Arms: 200 mg Mavoglurant
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this alcohol-interaction pilot study is to provide information on the effect of mavoglurant on the pharmacokinetics of alcohol and on alcohol responses, including stimulation, sedation, intoxication, body sway and physiological responses. The investigators propose to test the effects of 200 mg mavoglurant versus placebo on alcohol related responses. This is a between subjects double blind randomized design in which the investigators plan to run 40 subjects to obtain 28 completers.

DETAILED DESCRIPTION:
The purpose of this alcohol-interaction pilot study is to provide information on the effect of mavoglurant on the pharmacokinetics of alcohol and on alcohol responses, including stimulation, sedation, intoxication, body sway and physiological responses. The investigators propose to test the effects of 200 mg mavoglurant versus placebo on alcohol related responses. This is a between subjects double blind randomized design in which the investigators plan to run 40 subjects to obtain 28 completers.

Subjects will participate in two lab sessions, one prior to taking medication and one following 7-10 days of mavoglurant/placebo. During each session, participants will receive successive doses of alcohol over a 90 min period designed to raise their blood alcohol levels to 80 mg/dl; this dose was chosen because this is close to the legal limit of intoxication and to the peak BAC the investigators have observed in prior research studies. Subjects will be monitored throughout the lab session and will receive a phone call two days following the 2nd lab session and a follow-up appointment one week after the 2nd lab session to assess any remaining side effects from the medication.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 21-50
2. Able to read English at 6th grade level or higher and to complete study evaluations
3. Social drinkers
4. Willing to abstain from drinking alcohol during the outpatient study medication treatment period

Exclusion Criteria:

1. Seeking treatment for alcohol drinking
2. Current DSM-V criteria for any other substances, other than alcohol or nicotine.
3. Positive test results at any appointments after the initial intake appointment on urine drug screens conducted for opiates, cocaine, marijuana, benzodiazepines and/or barbiturates.
4. Regular use of psychoactive drugs including anxiolytics and antidepressants.
5. Psychotic or otherwise severely psychiatrically disabled.
6. Any medical conditions (including hepatic and renal impairment) that would contraindicate the consumption of alcohol or administration of mavoglurant.
7. History of neurological trauma or disease, delirium, or hallucinations, or any significant systemic illness or unstable medical condition.
8. Women who are pregnant, nursing, or refuse to use a reliable method of birth control. Urine pregnancy tests will be completed at intake and prior to administration of alcohol at each lab session.
9. Subjects who report disliking spirits will be excluded because hard liquor will be provided during the alcohol administration.
10. Subjects who have taken any investigational drug and/or participated in another study which involves additive blood sampling and/or interventional measures that would be considered excessive in combination with the current protocol within 4 weeks immediately preceding admission to the treatment period.
11. Subjects who report any daily drug use during the 30 days prior to randomization for the following: anxiolytics, beta blockers, central nervous system stimulants, hypnotics, non-therapeutic doses of neuroleptics and antidepressants, drugs with psychotropic activity or drugs which cause excessive sedation.
12. Subjects who have donated blood within the past six weeks.
13. Current use (within 30 days of screening) of specific psychoactive medications (e.g., typical neuroleptics, narcotic analgesics, antiparkinsonian medications, systemic corticosteroids, or medications with significant central anticholinergic activity, etc
14. Current use of warfarin.
15. Use of any medications that are contraindicated with mavoglurant and alcohol.
16. AST, ALT, total bilirubin >1.5 times upper normal; serum creatinine, >2 times upper normal limit, total bilirubin>1.5 times ULN; Serum creatinine >2.0 times ULN.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2023-07-13 (Actual); Study Completion 2023-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suchitra Krishnan-Sarin, PhD, Principal Investigator — Professor of Psychiatry
Locations (1):
- CMHC, Substance Abuse Center, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 34 Participants enrolled in the study, however there was an error in calculating alcohol dose in one participant. Analysis excluded this one participant, 33 analyzed at baseline.
  24 completed study and had outcome data, excluding this 1 participant, the final analysis is n=23.
Period: Overall Study
Arm/Group | 200 mg Mavoglurant | Placebo
Started | 17 | 17
Completed | 10 | 14
Not Completed | 7 | 3
Not completed — Adverse Event | 4 | 0
Not completed — Family/Personal issues | 3 | 2
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: 1 participant from the Mavoglurant condition was not included in the analysis due to an error in calculating alcohol dose (17 were randomized into that condition, 16 were analyzed).
Groups:
- Total: Total of all reporting groups
Arm/Group | 200 mg Mavoglurant | Placebo | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 17 | 33
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.3 (4.51) | 29.1 (6.68) | 27.7 (5.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 9 | 10 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 10
  Not Hispanic or Latino | 12 | 11 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 10 | 7 | 17
  Asian | 4 | 4 | 8
  Black | 1 | 2 | 3
  Multi-Race | 1 | 2 | 3
  Other | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 16 | 17 | 33

OUTCOME MEASURES:

1. Primary Outcome: Abnormal Labs and Adverse Events
Description: Number of participants (at Day 10; after both alcohol sessions and completed course of mavoglurant) with abnormal lab values or adverse events related to the interaction of alcohol and mavoglurant
Time Frame: Day 10
Population: 34 Participants enrolled in the study, however there was an error in calculating alcohol dose in one participant. Analysis excluded this one participant, 33 analyzed at baseline.
  24 completed study and had outcome data, excluding this 1 participant, the final analysis is n=23.
Measure: Count of Participants; unit: Participants
Arm/Group | 200 mg Mavoglurant | Placebo
Number analyzed (Participants) | 9 | 14
Participants
  Number of participants that reported Adverse Event(s) | 9 | 8
  Abnormal/Clinically Significant lab values after Mavoglurant and alcohol administration | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the course of the study from randomization to the 1 week follow-up visit; approximately 3 weeks.
Description: Standard definitions were used. The SAFTEE was utilized, this is a tool for systematic assessment of AE's which includes 1) open-ended questions about any changes in physical/health problems, appearance, or activity level, and 2) yes/no responses to a specific list of symptoms (typically associated with the Investigational Product).
Arm/Group | 200 mg Mavoglurant | Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 17/17 | 8/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 200 mg Mavoglurant (N=17) | Placebo (N=17)
Racing Heart (Cardiac disorders) | 1 (1) | 0 (0)
Mania/Hyperactivity (Psychiatric disorders) | 3 (3) | 0 (0)
Dissociation (Nervous system disorders) | 1 (1) | 0 (0)
Appetite Change (Gastrointestinal disorders) | 4 (4) | 0 (0)
Acid Indigestion (Gastrointestinal disorders) | 1 (2) | 0 (0)
Sore Arm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — From IV placement during study lab session
Back Ache (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 9 (10) | 1 (1)
Confusion (Nervous system disorders) | 2 (3) | 0 (0)
Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Extra sense of focus (Nervous system disorders) | 2 (2) | 0 (0)
Face Numbness (Nervous system disorders) | 1 (2) | 0 (0)
Fatigue (Nervous system disorders) | 2 (2) | 3 (3)
Feeling High/Intoxicated (Psychiatric disorders) | 3 (3) | 0 (0)
Frequent Urination (Renal and urinary disorders) | 0 (0) | 1 (2)
Good Mood / Awake (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 5 (6) | 2 (2)
Hurt Ankle (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Insomnia (Nervous system disorders) | 6 (8) | 2 (4)
Irritable (Psychiatric disorders) | 0 (0) | 1 (1)
Itchy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Lack of Focus (Nervous system disorders) | 4 (4) | 0 (0)
Memory Loss (Nervous system disorders) | 1 (1) | 0 (0)
Mood Altered (Psychiatric disorders) | 1 (1) | 0 (0)
Mouth and Throat Pain (General disorders) | 1 (2) | 0 (0)
Moving/Walking Slower (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle Twitch (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (6) | 4 (5)
Nervousness / Anxiety (Psychiatric disorders) | 6 (7) | 0 (0)
Night Sweats (Nervous system disorders) | 1 (1) | 0 (0)
Nightmares (Psychiatric disorders) | 1 (1) | 0 (0)
Pimples/Face Swelling (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sad (Psychiatric disorders) | 0 (0) | 1 (1)
Social Anxiety (Social circumstances) | 1 (1) | 0 (0)
Strange Feeling Behind the Eyes (Eye disorders) | 1 (1) | 0 (0)
Vision Felt Slower (Eye disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2)
Warm Feeling in Heart; the Feeling of God (General disorders) | 1 (1) | 0 (0)
Lightheaded (Nervous system disorders) | 3 (3) | 1 (1)
Saw Scary Faces While Sleeping (Nervous system disorders) | 0 (0) | 1 (1)
Sinus Pressure (General disorders) | 1 (1) | 0 (0)
Closer things looked closer; Farther things looked farther away (Eye disorders) | 1 (1) | 0 (0)
Hazy Vision (Eye disorders) | 0 (0) | 1 (1)
Trailing Vision (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-22): https://cdn.clinicaltrials.gov/large-docs/92/NCT03327792/Prot_SAP_001.pdf
  • Informed Consent Form (2023-06-30): https://cdn.clinicaltrials.gov/large-docs/92/NCT03327792/ICF_000.pdf